CLINICAL TRIAL: NCT03292367
Title: The Procedural Success and Complication Rate of the Left Distal Radial Approach for Coronary Angiography and Percutaneous Coronary Intervention. Prospective Observational Study
Brief Title: The Procedural Success and Complication Rate of the Left Distal Radial Approach
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seung Hwan Lee, Professor, Wonju Severance Christian Hospital
Other Study IDs: LeDRA
Record Dates: First submitted 2017-09-17; First posted 2017-09-25 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Radial Artery Injury at Wrist and Hand Level
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ldTRA: Patients who are planned to perform coronary angiography will be enrolled via left distal radial artery
  Interventions: Procedure: ldTRA

INTERVENTIONS:
Procedure: ldTRA — After puncture of left distal radial artery, coronary angiography and percutaneous coronary intervention, if needed, will be performed.

SUMMARY:
Left distal transradial approach (ldTRA) can be an attractive alternative route for left radial and right radial artery. Recently, Ferdinand Kiemeneij reported the feasibility and safety of the use of ldTRA. But, there is few studies focused on this issue. Therefore, the purpose of this prospective observational study is to assess the feasibility and safety of the ldTRA for CAG and PCI.

DETAILED DESCRIPTION:
Femoral artery has been traditionally used as a standard route for coronary angiography (CAG) and percutaneous coronary intervention (PCI). Recently, the frequency of use of transradial approach (TRA) is increasing. TRA has several advantages in terms of more comfortable feeling, immediate ambulation, less bleeding complication and decreased mortality rate compared to transfemoral approach (TFA). 2015 ESC guidelines recommend to use of radial artery in order to reduce bleeding complication and mortality. But, most operators tend to prefer right radial approach (RRA) for the access route, because they are usually right-handed and feel more comfortable in the use of right radial artery. Particularly when the patient is obese or the operator's height is short or has a herniated disc on neck or waist, the discomfort may become greater.

In other hand, left radial approach (LRA) have several advantages. Left brachial artery or subclavian artery is less tortuous than right side. The manipulation of catheter is similar with femoral approach. Also, since most patients are right-handed, compression after LRA leads to greater comfort for the patient.

In comparison to the convenience of the patient and procedure, comparative studies on clinical outcomes showed similar results for both RRA and LRA. But LRA may be more at risk for radiation. This is because the operator has to lean more toward the patient for the procedure, which can result in increased radiation exposure.

Recently, the left distal radial artery approach (ldTRA) has been introduced as an alternative to feasibility and safety while satisfying both patient and operator convenience. The left palm is positioned facing the floor at the left groin. Left distal radial artery is punctured at the level of anatomical snuffbox. Ferdinand Kiemeneij reported that CAG and PCI were successfully performed in 70 patients.

There are no nerve and vein in the anatomical snuffbox. And distal radial artery is located at superficial area. So, there may be potential advantage to reduce bleeding complication and nerve injury. Moreover, ldTRA can be an alternative method for the patient requiring arteriovenous fistula and for the patient preparing coronary artery bypass graft because there is no injury of left radial artery.

The patients have potential bleeding risk because dual antiplatelet agents (aspirin 300mg and clopidogrel 300mg) and more than 3,000 units of unfractionated heparin should be loaded for CAG and PCI. The effective hemostasis method has not yet been established after ldTRA. Therefore, it is important to establish effective hemostasis method and timing. However, like TRA, ldTRA requires a learning curve to be mastered, and it cannot be performed if the pulse is not palpable. There are few studies related to ldTRA. The purpose of this prospective observational study is to assess the feasibility and safety of the ldTRA for CAG and PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years old requiring coronary angiography
* Patients who are palpable left distal radial artery
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who are not palpable left distal radial artery
* Patients who are positive in Modified Allen's test (suspicious of occlusion of ulnar artery)
* Pregnant women
* Patients who are not appropriate for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During 1 year, more than 200 patients who are needed to perform coronary angiography or percutaneous coronary intervention will be prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Success rate of coronary angiography | 1 year
  The frequency of success rate of coronary angiography (%)
Success rate of percutaneous coronary intervention | 1 year
  The frequency of success rate of percutaneous coronary intervention (%)

SECONDARY OUTCOMES:
Success rate of puncture of left distal radial artery | 1 year
  The frequency rate of successful puncture of left distal radial artery (%)
Diameter of left distal radial artery | 1 year
  Measured by ultrasonography before procedure (mm)
Hemostasis duration at the puncture site | 1 year
  Hemostasis duration after procedure (minute)
Complications at the puncture site | 1 year
  The frequency rate of complications at the puncture site (%)
Procedure time | 1 year
  Procedure time including coronary angiograph and percutaneous coronary intervention, if performed (minute)
Exposure time of radiation | 1 year
  Total exposure time of radiation during procedure (minute)
Dose of radiation | 1 year
  Dose of radiation during procedure (Gy-cm2)
The degree of patient's satisfaction | 1 year
  Questionnaire using visual analogue scale for the pain and satisfaction of overall procedure especially focused on the left distal radial approach (Maximum 10 score, Minimum 0 score)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Wonju Severance Christian Hospital, Yonsei University Wonju College of Medicine
Locations (1):
- Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941